CLINICAL TRIAL: NCT06544473
Title: Determining Dose Equivalence Between Oral and Transdermal Estrogen Treatment in Women With Turner Syndrome - A Randomized Study
Brief Title: Determining Dose Equivalence Between Oral and Transdermal Estrogen Treatment in Women With Turner Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AU2019TS1
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-07

CONDITIONS: Turner Syndrome; Hypogonadism; Ovarian; Hormone Replacement Therapy; Estrogen Replacement Therapy; Estrogen Deficiency
Keywords: Turner syndrome; Hormone Replacement Therapy; Estrogen Replacement Therapy; Estrogen treatment; Dose equipotency
MeSH Terms: conditions — Turner Syndrome; Hypogonadism | interventions — Estradiol; estradiol, estriol drug combination

STUDY DESIGN:
Intervention Model Description: A randomized crossover study
Masking Description: The patients with TS will be randomized to receive either oral (tablet) or transdermal (gel) estrogen replacement therapy. The study is not blinded, as both investigator and study participants know which medication, they are receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral estrogen treatment (Active Comparator): Turner syndrome patients receiving oral estrogen treatment (Estrofem®)
  Interventions: Drug: 17-beta estradiol
- Transdermal estrogen treatment (Active Comparator): Turner syndrome patients receiving transdermal estrogen treatment (Divigel)
  Interventions: Drug: 17-beta estradiol

INTERVENTIONS:
Drug: 17-beta estradiol — Treatment with orally administered estrogen for 14 days
  Other Names: Estrofem
  Arms: Oral estrogen treatment
Drug: 17-beta estradiol — Treatment with transdermally administered estrogen for 14 days
  Other Names: Divigel
  Arms: Transdermal estrogen treatment

SUMMARY:
This 5-week, phase IV randomized crossover trial aims to compare the effects of oral versus transdermal estrogen replacement therapy (ERT) in women with Turner syndrome (TS). The objective is to establish the equipotency between the two estradiol regimens by evaluating various estradiol-dependent surrogate markers. The study involves 50 women with TS, aged 18-50 years, who are randomized to receive either oral or transdermal ERT for 14 days, followed by a crossover to the alternate treatment for another 14 days, with a one-week washout period in between. Blood tests are conducted at baseline, after the first 14 days of treatment, after the washout period, and after the final 14 days of treatment. The investigators anticipate that this study will provide clinicians with a better understanding of ERT in treating women with TS.

DETAILED DESCRIPTION:
OBJECTIVE

1. To determine the equipotency of two different estradiol regimens (oral versus transdermal administration) using various estradiol-dependent surrogate markers.

BACKGROUND Turner syndrome (TS) is a rare genetic condition affecting approximately 1 in 2,000 female births. A hallmark of TS is ovarian dysgenesis, leading to hypogonadism, premature ovarian failure, and infertility. Consequently, estrogen replacement therapy (ERT) is typically initiated around age 11-12 to induce puberty and continued until the average age of menopause (50-55 years), aiming for at least 42 years of adequate estrogen exposure.

Hypogonadism in TS is associated with various health complications. Importantly, estradiol (E2) replacement may mitigate these risks. Estrogen deficiency in TS affects cardiovascular health (hypertension, congenital cardiac disease, altered lipid profiles), metabolic function (diabetes, thyroid dysfunction, hepatic disorders, kidney disease, skeletal abnormalities), and is linked to neurocognitive and social challenges.

E2 can be administered orally or transdermally (TD), but it remains unclear whether either route offers specific advantages. There is ongoing debate regarding a potential increased thromboembolic risk in TS patients treated with oral E2. Epidemiological studies in postmenopausal women have reported an elevated thromboembolic risk associated with oral estrogen treatment, but to a lesser extent with TD administration. However, extrapolating data from postmenopausal women to TS patients is inappropriate, as women with TS receive estrogen as replacement therapy due to inadequate endogenous production. Furthermore, limited knowledge exists regarding the side effects of oral versus TD estrogen replacement therapy for TS patients.

MATERIALS AND METHODS

Women aged 18-50 years with TS recruited primarily from the Department of Endocrinology at Aarhus University Hospital (n=50); 300 patients with TS are currently followed in the outpatient clinic. The investigators also have the opportunity to recruit from the Turner Association in Denmark, and finally the investigators do have contact with other outpatient clinics with TS patients in Denmark from where the investigators have previously recruited TS patients.

Design:

A 5-week, phase IV randomized crossover trial involving 50 women with TS. Participants are randomized to receive E2 for 14 days, either as oral or TD treatment, followed by a crossover to the alternate treatment for another 14 days, with a one-week washout period in between.

Laboratory analyses:

Blood samples are collected at baseline, after the first 14 days of treatment, after the washout period, and after the final 14 days of treatment.

STATISTICS

Data will be summarized by treatment group and assessment time point. The investigators will use a mixed model with repeated measures analysis of variance (ANOVA) to compare the mean changes in each of the study variables between treatments over time. When appropriate, transformations or nonparametric methods will be used. All tests are two-tailed with a 5% level of significance. Data are presented as mean ± SE or median with CI for metrics not normally distributed.

PERSPECTIVES

Patients with TS undergo hormone replacement therapy from puberty to menopause, spanning more than 40 years of treatment. To date, only two experimental studies have compared oral and TD ERT in TS, focusing solely on metabolic parameters and finding no differences between the two regimens. The investigators aim for this study to provide clinicians with a better understanding of ERT in treating women with TS, and to contribute with new knowledge about hormonal treatment for the general population as well.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of TS regardless of karyotype
* Age 18-50 years
* Already receiving estrogen treatment

Exclusion Criteria:

* Active systemic chronic diseases
* Known or suspected breast cancer
* Known or suspected estradiol-dependent tumors (endometrial cancer or similar)
* Untreated endometrial hyperplasia
* Current or previous venous thromboembolism
* Acute or previous liver disease where liver enzymes are still elevated by a factor 3 or more
* Known hypersensitivity to the medications used
* Pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only patients with Turner syndrome can participate
Enrollment: 50 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Equipotency | After 14 days
  Levels of luthenizing hormone and follicle stimulating hormone are measured at different doses

CONTACTS AND LOCATIONS:
Overall Officials: Claus H Gravholt, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stochholm K, Juul S, Juel K, Naeraa RW, Gravholt CH. Prevalence, incidence, diagnostic delay, and mortality in Turner syndrome. J Clin Endocrinol Metab. 2006 Oct;91(10):3897-902. doi: 10.1210/jc.2006-0558. Epub 2006 Jul 18. PMID 16849410
- [Background] Gravholt CH, Andersen NH, Conway GS, Dekkers OM, Geffner ME, Klein KO, Lin AE, Mauras N, Quigley CA, Rubin K, Sandberg DE, Sas TCJ, Silberbach M, Soderstrom-Anttila V, Stochholm K, van Alfen-van derVelden JA, Woelfle J, Backeljauw PF; International Turner Syndrome Consensus Group. Clinical practice guidelines for the care of girls and women with Turner syndrome: proceedings from the 2016 Cincinnati International Turner Syndrome Meeting. Eur J Endocrinol. 2017 Sep;177(3):G1-G70. doi: 10.1530/EJE-17-0430. PMID 28705803
- [Background] Hjerrild BE, Mortensen KH, Gravholt CH. Turner syndrome and clinical treatment. Br Med Bull. 2008;86:77-93. doi: 10.1093/bmb/ldn015. Epub 2008 Apr 9. PMID 18400842
- [Background] Gravholt CH, Landin-Wilhelmsen K, Stochholm K, Hjerrild BE, Ledet T, Djurhuus CB, Sylven L, Baandrup U, Kristensen BO, Christiansen JS. Clinical and epidemiological description of aortic dissection in Turner's syndrome. Cardiol Young. 2006 Oct;16(5):430-6. doi: 10.1017/S1047951106000928. PMID 16984695
- [Background] Mortensen KH, Andersen NH, Hjerrild BE, Horlyck A, Stochholm K, Hojbjerg Gravholt C. Carotid intima-media thickness is increased in Turner syndrome: multifactorial pathogenesis depending on age, blood pressure, cholesterol and oestrogen treatment. Clin Endocrinol (Oxf). 2012 Dec;77(6):844-51. doi: 10.1111/j.1365-2265.2012.04337.x. PMID 22233516
- [Background] Mauger C, Lancelot C, Roy A, Coutant R, Cantisano N, Le Gall D. Executive Functions in Children and Adolescents with Turner Syndrome: A Systematic Review and Meta-Analysis. Neuropsychol Rev. 2018 Jun;28(2):188-215. doi: 10.1007/s11065-018-9372-x. Epub 2018 Apr 27. PMID 29704077
- [Background] Hansen M. Female hormones: do they influence muscle and tendon protein metabolism? Proc Nutr Soc. 2018 Feb;77(1):32-41. doi: 10.1017/S0029665117001951. Epub 2017 Aug 29. PMID 28847313
- [Background] Greising SM, Baltgalvis KA, Lowe DA, Warren GL. Hormone therapy and skeletal muscle strength: a meta-analysis. J Gerontol A Biol Sci Med Sci. 2009 Oct;64(10):1071-81. doi: 10.1093/gerona/glp082. Epub 2009 Jun 26. PMID 19561145
- [Background] Canonico M, Plu-Bureau G, Lowe GD, Scarabin PY. Hormone replacement therapy and risk of venous thromboembolism in postmenopausal women: systematic review and meta-analysis. BMJ. 2008 May 31;336(7655):1227-31. doi: 10.1136/bmj.39555.441944.BE. Epub 2008 May 20. PMID 18495631
- [Background] Renoux C, Dell'aniello S, Garbe E, Suissa S. Transdermal and oral hormone replacement therapy and the risk of stroke: a nested case-control study. BMJ. 2010 Jun 3;340:c2519. doi: 10.1136/bmj.c2519. PMID 20525678
- [Background] Sweetland S, Beral V, Balkwill A, Liu B, Benson VS, Canonico M, Green J, Reeves GK; Million Women Study Collaborators. Venous thromboembolism risk in relation to use of different types of postmenopausal hormone therapy in a large prospective study. J Thromb Haemost. 2012 Nov;10(11):2277-86. doi: 10.1111/j.1538-7836.2012.04919.x. PMID 22963114
- [Background] Gravholt CH, Naeraa RW, Fisker S, Christiansen JS. Body composition and physical fitness are major determinants of the growth hormone-insulin-like growth factor axis aberrations in adult Turner's syndrome, with important modulations by treatment with 17 beta-estradiol. J Clin Endocrinol Metab. 1997 Aug;82(8):2570-7. doi: 10.1210/jcem.82.8.4127. PMID 9253336
- [Background] Taboada M, Santen R, Lima J, Hossain J, Singh R, Klein KO, Mauras N. Pharmacokinetics and pharmacodynamics of oral and transdermal 17beta estradiol in girls with Turner syndrome. J Clin Endocrinol Metab. 2011 Nov;96(11):3502-10. doi: 10.1210/jc.2011-1449. Epub 2011 Aug 31. PMID 21880799
- [Background] Torres-Santiago L, Mericq V, Taboada M, Unanue N, Klein KO, Singh R, Hossain J, Santen RJ, Ross JL, Mauras N. Metabolic effects of oral versus transdermal 17beta-estradiol (E(2)): a randomized clinical trial in girls with Turner syndrome. J Clin Endocrinol Metab. 2013 Jul;98(7):2716-24. doi: 10.1210/jc.2012-4243. Epub 2013 May 15. PMID 23678038
- [Background] Gravholt CH, Naeraa RW, Nyholm B, Gerdes LU, Christiansen E, Schmitz O, Christiansen JS. Glucose metabolism, lipid metabolism, and cardiovascular risk factors in adult Turner's syndrome. The impact of sex hormone replacement. Diabetes Care. 1998 Jul;21(7):1062-70. doi: 10.2337/diacare.21.7.1062. PMID 9653596
- [Background] Klein KO, Baron J, Colli MJ, McDonnell DP, Cutler GB Jr. Estrogen levels in childhood determined by an ultrasensitive recombinant cell bioassay. J Clin Invest. 1994 Dec;94(6):2475-80. doi: 10.1172/JCI117616. PMID 7989605
- [Background] Klein KO, Rosenfield RL, Santen RJ, Gawlik AM, Backeljauw PF, Gravholt CH, Sas TCJ, Mauras N. Estrogen Replacement in Turner Syndrome: Literature Review and Practical Considerations. J Clin Endocrinol Metab. 2018 May 1;103(5):1790-1803. doi: 10.1210/jc.2017-02183. PMID 29438552
- [Background] Berglund A, Stochholm K, Gravholt CH. The epidemiology of sex chromosome abnormalities. Am J Med Genet C Semin Med Genet. 2020 Jun;184(2):202-215. doi: 10.1002/ajmg.c.31805. Epub 2020 Jun 7. PMID 32506765